CLINICAL TRIAL: NCT07046975
Title: Bioavailability and Bioequivalence (BA/BE) Study of Extended Release (ER) Torsemide and Spironolactone Fixed Dose Combination (FDC) Tablet in Healthy Adult Human Subjects
Brief Title: Bioavailability and Bioequivalence Study of Extended Release Torsemide and Spironolactone
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAR-HS-027-24
Record Dates: First submitted 2025-06-06; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Bioavailability Heathy Volunteers
Keywords: Torsemide; Spironolactone; Combination; Bioavailability
MeSH Terms: interventions — Torsemide; Spironolactone

STUDY DESIGN:
Intervention Model Description: Open label, randomized, two-period, two-sequence, balanced, multiple-dose crossover intrasubject variability and steady-state BA/BE study
Masking Description: The study is of randomized open label design; as it is not essential to design the study as double-blind for assessing bioavailability of formulations. The analyst will not have access to the randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 FDC (Active Comparator): Fixed Dose Combination (FDC) 12 mg ER Torsemide and 15 mg Spironolactone tablet
  Interventions: Drug: Torsemide and Spironolactone tablet; Drug: Torsemide Tablets and Spironolactone Tablets
- Arm 2 (Torsemide tablets and Spironolactone tablets) (Active Comparator): 10 mg Torsemide and 25 mg Spironolactone tablets given together
  Interventions: Drug: Torsemide and Spironolactone tablet; Drug: Torsemide Tablets and Spironolactone Tablets

INTERVENTIONS:
Drug: Torsemide and Spironolactone tablet — Fixed Dose Combination (FDC): (12 mg Extended Release (ER) Torsemide and 15 mg Spironolactone) tablet
Drug: Torsemide Tablets and Spironolactone Tablets — 10 mg Torsemide tablet and 25 mg Spironolactone tablet given together

SUMMARY:
To study intrasubject variability and steady-state pharmacokinetics of multiple-doses of Extended Release Torsemide and Spironolactone Fixed Dose Combination (FDC) tablets given together in healthy adult subjects.

DETAILED DESCRIPTION:
To study intrasubject variability and steady-state pharmacokinetics of the multiple-doses of Extended Release (ER) Torsemide and Spironolactone Fixed Dose Combination (FDC) (12 mg ER Torsemide and 15 mg Spironolactone) tablet and 10 mg Torsemide and 25 mg Aldactone® (Spironolactone) tablets given together in healthy adult subjects. In addition, torsemide, sodium, potassium, and creatinine will be measured in the urine samples.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

1. Healthy human adult subjects within the age range of 18 to 45 years [both inclusive].
2. Weight not less than 50 kg for male and 45 kg for female and BMI 18.50 to 29.99 kg/m2 [both inclusive].
3. Willingness to provide written informed consent to participate in the study.
4. Subjects should be non-smoker [defined as someone who has stopped smoking for a year before the date of screening] and should not be consuming tobacco containing products.
5. Free of significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
6. Absence of disease markers of HIV 1 and 2, Hepatitis B and C and Syphilis.
7. Subject should be literate.
8. Male subjects must be using two acceptable methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the study, and upto the study completion visit. Subjects must refrain from fathering a child in the next two weeks following the last study drug administration or have undergone vasectomy (vasectomy must have been done more than 6 months prior to first dosing). Contraceptive usage requirement will be conveyed during the inform consent process. Subjects will be advised to follow effective method of contraception until 2 weeks after the last dose is given.
9. Female subjects of childbearing potential must be using two acceptable methods of contraception, (e.g., intra-uterine device (IUD) plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the study and for two weeks following the last study drug administration. Contraceptive usage requirement will be conveyed during the inform consent process (or) Postmenopausal women for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy have been performed).

Exclusion Criteria:

Any of the following conditions are cause for exclusion from the study:

1. History or presence of significant: cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, musculoskeletal, psychiatric disease/disorder.
2. History or presence of significance:

   Asthma, urticaria, or other allergic-type reactions after taking Torsemide, Spironolactone or any other drug.

   Ulceration or history of gastric and/or duodenal ulcer. Stomach or intestinal bleeding. Jaundice in the past 6 months. Internal bleeding.
3. Hypersensitivity or allergy to Torsemide, Spironolactone or any of the excipients.
4. History of alcohol or drug abuse in the past one year.
5. Family history of bleeding disorders.
6. History of difficulty in passing urine or emptying the bladder or of incontinence.
7. Have donated 500 mL or more blood within 90 days before receiving the first dose of the study drug.
8. Subjects who have participated in another clinical study in the past 3 months prior to commencement of this study.
9. Any difficulty in the accessibility of forearm veins for cannulation or blood sampling and or difficulty with donating blood.
10. Refuse to abstain from food for at least 10 h prior to dosing and for at least 4 h after dosing in each period.
11. Refuse to abstain from fluid for at least 1 h before and 1 h after dosing in each period (except 240 ± 2 mL water given for dosing).
12. Found positive during breath alcohol test done during period one check-in and inability to abstain from alcohol till the end of the study.
13. Found positive during urine drug screening done prior to period one check-in.
14. Found positive screening results for Hepatitis B, Hepatitis C, HIV, or Syphilis.
15. History of difficulty in swallowing tablets.
16. Received any medication [including over-the-counter products], herbal products for 14 days preceding the study.
17. Use of enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
18. History of dehydration from diarrhea, vomiting, or any other reason within 24 hours prior to check-in of period one.
19. Consumption of xanthine-containing food and beverages (chocolates, tea, coffee, or cola drinks) for at least 48 hours prior to check-in of period one.
20. Consumption of grapefruit or its products within the 48 hours prior to check-in of period one.
21. Female subjects are found to be positive during pregnancy tests done prior to period one check-in.
22. Lactating females.
23. Investigator/Physician feels that it is not in the subject's and/or study's best interest to enroll the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Plasma (Blood) sample analysis of torsemide for Cmax | 24 hours
  Measurement of torsemide in the blood for Cmax.
Plasma (Blood) sample analysis of torsemide for AUC | 24 hours
  Measurement of torsemide in the blood for AUC.
Plasma (Blood) sample analysis of Spironolactone and Canrenone for Cmax | 24 hours
  Measurement of Spironolactone and Canrenone in the blood (Active metabolite of spironolactone) for Cmax.
Plasma (Blood) sample analysis of AUC in the blood for Spironolactone and Canrenone | 24 hours
  Measurement of Spironolactone and Canrenone (Active metabolite of spironolactone) for AUC.
Urine sample analysis to determine urinary excretion | 24 hours
  Urine samples will be used to calculate urinary excretion at each timepoint and the total in 24 hours.
Urine sample analysis for torsemide secretion | 24 hours
  Calculate percentage of torsemide recovered in the urine.
Urine sample analysis of torsemide for Rmax | 24 hours
  Urinary torsemide excretion will be measured for Rmax.
Urine sample analysis for electrolytes | 24 hours
  Electrolytes (sodium, potassium) will be measured to determine the percentage of drug recovered.
Urine sample analysis for creatinine | 24 hours
  Urinary creatinine will be measured at each timepoint over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Shah, PhD, JD, Study Director — Sarfez Pharmaceuticals, Inc.
Locations (1):
- Sarfez Pharmaceuticals, Vienna, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
HIPAA